CLINICAL TRIAL: NCT05029219
Title: A Prospective Randomized Controlled Study for the Efficacy of Virtual Reality Intervention Procedure Simulator on the Training of Pain Procedures
Brief Title: Virtual Reality Intervention Procedure Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeong Kim, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3-2021-0237
Record Dates: First submitted 2021-08-11; First posted 2021-08-31 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Novice Doctor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): To become proficient in lumbar transforaminal epidural blocks, participants receive additional training using virtual reality programs after audiovisual education.
  Interventions: Device: Arm I (Virtual reality group)
- Self study group (Active Comparator): In order to become proficient in lumbar transforaminal epidural block, participants have self-study time using books and videos after audiovisual education.
  Interventions: Device: Arm II (Self study group)

INTERVENTIONS:
Device: Arm I (Virtual reality group) — In the preparatory session, the participant is given a survey. It is about demographic information such as gender, age, and age, as well as prior experience with the procedure. The primary test is performed with a fluoroscopy guided lumbar transforaminal epidural block with a human-shaped phantom.
  After that, the test group and the control group receive the same audiovisual education for about 5 minutes. The test group receives about 60 minutes of training using a virtual reality program.
  Arms: Virtual reality group
Device: Arm II (Self study group) — In the preparatory session, the participant is given a survey. It is about demographic information such as gender, age, and age, as well as prior experience with the procedure. The primary test is performed with a fluoroscopy guided lumbar transforaminal epidural block with a human-shaped phantom.
  After that, the test group and the control group receive the same audiovisual education for about 5 minutes. The control group have provided with video materials and books provided during audiovisual education and have given time for self-study for 60 minutes. Subsequently, a second test is performed with a fluroscopy-guided lumbar transforaminal epidural block with a human-shaped phantom.
  Arms: Self study group

SUMMARY:
The purpose of this study is to prove the effectiveness of the virtual reality program in educating lumbar transforaminal epidural blocks to novice doctors.

ELIGIBILITY:
Inclusion Criteria:

* Residents in department of anesthesiology and pain medicine unfamiliar with fluoroscopy guided epidural block

Exclusion Criteria:

* Residents in department of anesthesiology and pain medicine familiar with fluoroscopy guided epidural block

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Checklist score | 60 min of education programs
  When all training courses are completed and a post-test is performed on the phantom, it is determined how much the checklist score has changed compared to the screening time.
  Range from 0 to 7. Minimum score means worst and maximum score means good performance.

SECONDARY OUTCOMES:
Global rating score | 60 min of education programs
  When all training courses are completed and a post-test is performed on the phantom, it is determined how much the global rating score has changed compared to the screening time.
  Range from 7 to 35. Minimum score means worst and maximum score means good performance.
Time taken to perform lumbar transforaminal epidural injection | Procedure duration
  During the pre-test and post-test, how long it takes to perform the procedure is compared.
Number of fluroscopy shots when performing lumbar transforaminal epidural injection under a fluoroscopy guide | Procedure duration
  It is determined by comparing the number of fluroscopy pictures
Participants' satisfaction with the curriculum | 60 min of education programs
  After the completion of all training and testing sessions, have participants rate their satisfaction with the training on a 100-point scale.
  Range from 0 to 100. Minimum score means less satisfaction and maximum score means better satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea